CLINICAL TRIAL: NCT04851275
Title: Increasing Decision Quality in Older Men in Selecting Treatment Options for Lower Urinary Tract Symptoms (LUTS): A Pilot Randomized Controlled Trial
Brief Title: Increasing Decision Quality for Men With Lower Urinary Tract Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SingHealth Polyclinics (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2018/3106
Record Dates: First submitted 2021-03-26; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Patient Engagement; Patient Preference
MeSH Terms: conditions — Patient Participation; Patient Preference

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared decision making for men with lower urinary tract symptoms (Experimental): Participants used the Visual Analogue Uroflowmetry Score so report their symptoms and were attended by Primary Care Physicians trained in shared decision making
  Interventions: Behavioral: Physicians trained in shared decision making
- No shared decision making for men with lower urinary tract symptoms (Active Comparator): Participants did not use the Visual Analogue Uroflowmetry Score to report their symptoms and received usual care by Primary Care Physicians not trained in shared decision making
  Interventions: Behavioral: Physicians were not trained in shared decision making

INTERVENTIONS:
Behavioral: Physicians trained in shared decision making — Physicians in this group were trained in shared decision making
  Arms: Shared decision making for men with lower urinary tract symptoms
Behavioral: Physicians were not trained in shared decision making — Physicians did not receive training in shared decision making
  Arms: No shared decision making for men with lower urinary tract symptoms

SUMMARY:
In this study, the investigators show that by upskilling of primary care physicians (PCPs) in SDM and leveraging on a novel pictorial Visual Analogue Uroflowmetry Score (VAUS), they can enhance older men's recognition of LUTS and stimulated discussion with their PCPs.

DETAILED DESCRIPTION:
Lower urinary tract symptoms (LUTS), often related to prostatomegaly, is common but seldom sought medical attention amongst older men. Visual-aid and shared decision-making (SDM) are potential solutions to address LUTS. The study aimed to determine the effect of a novel pictorial Visual Analogue Uroflowmetry Score (VAUS) and primary care physicians (PCP) SDM training on the decisional quality amongst men selecting their treatment options for LUTS.

This study recruited 60 multi-ethnic Asian men aged ≥50 years with moderate-to-severe LUTS (International Prostate Symptoms Score≥8 and/or QOL≥3) in a Singapore public primary care clinic. Men used the VAUS to report their symptoms. 60 men were randomly assigned to PCPs trained in SDM in the intervention group (n=30) and the other 30 to the control group (PCPs without SDM-training). Patient-physician dyad decision quality was measured using the validated SDMQ-9 (patient) and SDMQ-Doc (physician) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* men aged 50 years old and older attending the polyclinic for routine follow up of a chronic disease (non-communicable disease)
* have moderate-to-severe LUTS and/or poor quality of life (QOL) as assessed by the validated International Prostate Symptom Score (IPSS) of eight or more and/or its individual QOL score of three or more
* men of any local Asian ethnicity and were willing to provide written consent
* can communicate with their allocated PCP in either of the three main local languages; English, Mandarin or Malay.

Exclusion Criteria:

* have indwelling catheters
* urinary incontinence requiring diapers
* anuria due to any renal pathology
* gross hematuria
* acute urinary retention
* symptoms consistent with an acute urinary tract infection
* existing treatment of LUTS or other prostate pathology
* visual or hearing impairment which render men incapable of understanding the study procedure and providing informed consent
* men unwilling to discuss their LUTS treatment options with their PCP

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Quality of the decision on the management of lower urinary tract symptoms from the patients' perspective | Through study completion, an average of 6 months
  The Shared Decision Making-9 (SDMQ9) Questionnaire measures decision quality from the perspective of the patient. Nine individual items in the questionnaire is scored from 0 to 5 on a six-point Likert scale ranging from 0 ("completely disagree") to 5 ("completely agree"). Standard scoring for the full scale is the total score, with values from 0 to 45. Higher scores indicate higher quality decisions.
Quality of the decision on the management of lower urinary tract symptoms from the physicians' perspective | Through study completion, an average of 6 months
  The Shared Decision Making-Doctor (SDMQDoc) Questionnaire measures decision quality from the perspective of the physician. Nine individual items in the questionnaire is scored from 0 to 5 on a six-point Likert scale ranging from 0 ("completely disagree") to 5 ("completely agree"). Standard scoring for the full scale is the total score, with values from 0 to 45. Higher scores indicate higher quality decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Tan Ngiap Chuan, MBBS, Study Director — Singhealth polyclinic
Locations (1):
- Haidee Ngu, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tiwari R, Ng MY, Neo SH, Mangat R, Ho H. Prospective validation of a novel visual analogue uroflowmetry score (VAUS) in 1000 men with lower urinary tract symptoms (LUTS). World J Urol. 2020 May;38(5):1267-1273. doi: 10.1007/s00345-019-02909-1. Epub 2019 Aug 27. PMID 31451932